CLINICAL TRIAL: NCT06317051
Title: A Phase III/IV Factorial Randomized Double-blind Trial to Compare the Addition of Dapagliflozin vs Placebo and Rosuvastatin/Ezetimibe Versus Pitavastatin in Patients With HIV on Integrase Strand Transfer Inhibitor-based Antiretrovirals With Elevated Metabolic Risk
Brief Title: Optimising Metabolic Management for People With Human Immunodeficiency Virus (HIV) on Integrase Based Antiretroviral Therapy (ART)
Acronym: OPTIMAR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: OPTIMAR
Record Dates: First submitted 2024-02-21; First posted 2024-03-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Weight Gain
Keywords: HIV
MeSH Terms: conditions — HIV Infections; Weight Gain | interventions — dapagliflozin; pitavastatin; Tablets; Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dapagliflozin 10mg + pitavastatin 4mg (Active Comparator): Dapagliflozin 10mg + pitavastatin 4mg given as daily tablets for 48 weeks
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Pitavastatin 4 Mg Oral Tablet
- Dapagliflozin 10mg + rosuvastatin 10mg/ezetimibe 10mg (Active Comparator): Dapagliflozin 10mg + rosuvastatin 10mg/ezetimibe 10mg given as daily tablets for 48 weeks
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Rosuvastatin and Ezetimibe
- Placebo + pitavastatin 4mg (Placebo Comparator): Placebo + pitavastatin 4mg given as daily tablets for 48 weeks
  Interventions: Drug: Pitavastatin 4 Mg Oral Tablet; Drug: Placebo
- Placebo + rosuvastatin 10mg/ezetimibe 10mg (Placebo Comparator): Placebo + rosuvastatin 10mg/ezetimibe 10mg given as daily tablets for 48 weeks
  Interventions: Drug: Rosuvastatin and Ezetimibe; Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin will be administered as a comparator to the placebo to assess its effects on weight reduction
  Other Names: FORXIGA
  Arms: Dapagliflozin 10mg + pitavastatin 4mg; Dapagliflozin 10mg + rosuvastatin 10mg/ezetimibe 10mg
Drug: Pitavastatin 4 Mg Oral Tablet — Pitavastatin tablets will be administered as a comparator to Rosuvastatin/Ezetimibe 10mg/10mg tablets to assess and compare their effects on LDL concentrations
  Other Names: Livazo
  Arms: Dapagliflozin 10mg + pitavastatin 4mg; Placebo + pitavastatin 4mg
Drug: Rosuvastatin and Ezetimibe — Rosuvastatin/Ezetimibe 10mg/10mg tablets will be administered as a comparator to pitavastatin to assess and compare their effects on LDL concentrations
  Arms: Dapagliflozin 10mg + rosuvastatin 10mg/ezetimibe 10mg; Placebo + rosuvastatin 10mg/ezetimibe 10mg
Drug: Placebo — The placebo tablets are visually identical to the active drug tablets and will be administered as a comparator to Dapagliflozin.
  Arms: Placebo + pitavastatin 4mg; Placebo + rosuvastatin 10mg/ezetimibe 10mg

SUMMARY:
People with HIV are at a higher risk of cardiovascular diseases (CVD) due to the effects of the virus and its treatment. Integrase strand transfer inhibitors (INSTIs), a common HIV treatment, are associated with increased CVD risk and metabolic issues, such as weight gain and high blood pressure. Sodium-glucose cotransporter 2 (SGLT2) inhibitors, however, have been working well in reducing CVD events and hospitalizations due to heart failure, irrespective of diabetes presence. They also help in reducing weight and blood pressure. Pitavastatin has shown to work in lowering CVD events in people with HIV, but its availability is limited. This benefit is thought to be common to all statins, but this has not yet been confirmed. This study will examine the impact of dapagliflozin vs. placebo on metabolic parameters in people with HIV with high metabolic risk who are on INSTI-based ART.

DETAILED DESCRIPTION:
This is a 2x2 factorial, randomised, placebo-controlled, double-blind, phase III/IV trial with two randomisations performed centrally via an on-line system, stratified by site. Participants will be randomised 1:1 to dapagliflozin 10mg vs. Placebo; this randomisation will be blinded. Participants will also be randomised 1:1 within each group to pitavastatin 4mg vs. rosuvastatin 10mg/ezetimibe 10mg; this randomisation will be open label.

Therefore, participants will be randomised to one of 4 groups:

1. Dapagliflozin 10mg + pitavastatin 4mg
2. Dapagliflozin 10mg + rosuvastatin 10mg/ezetimibe 10mg
3. Placebo + pitavastatin 4mg
4. Placebo + rosuvastatin 10mg/ezetimibe 10mg

With the following 2-arm randomised comparisons:

* Primary analysis hypothesis: a+b vs c+d (dapagliflozin vs placebo)
* Secondary analysis hypothesis: a+c vs b+d (pitavastatin vs rosuvastatin 10mg/ezetimibe 10mg)

The study's primary and secondary endpoints described will assess both efficacy and safety/tolerability across randomisation arms. Follow up will continue to 48 weeks and endpoint measures will be obtained at 4, 12, 24, and 48 weeks. Primary endpoint is at 24 weeks. The total number of participants is 300, with 75 randomised to each of the groups as listed above.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years and at least one of the following risk factors:

   1. BMI > 7% increase or > 5kg weight gain since INSTI commencement, or
   2. BMI ≥ 30 kg/m2
2. BMI ≥18 kg/m2 prior to INSTI commencement
3. Currently taking INSTI-based ART
4. Sustained virologic response, defined as viral load <200 copies/mL for at least 12 months
5. Current CD4 >250 cells/mm3
6. Informed consent for trial participation

Exclusion Criteria:

1. Currently taking a protease inhibitor
2. Indicated to take or already taking high intensity statin
3. estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
4. Currently taking an SGLT-2 inhibitor or glucagon-like peptide 1 (GLP-1) agonist
5. Absolute contraindication or absolute indication to SGLT2 inhibitor therapy
6. Absolute contraindication to pitavastatin, rosuvastatin, ezetimibe or combination of rosuvastatin/ezetimibe
7. Pregnant or breast feeding
8. Severe hepatic impairment (Child Pugh B or C)
9. Participants receiving any excluded/contraindicated medication
10. Participants who are enrolled into an additional interventional study.
11. Expected inability or unwillingness to participate in study procedures.
12. In the opinion of the investigator, participation in a trial is not in the best interest of the patient.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of dapagliflozin vs. placebo on weight reduction | 24 weeks
  Mean reduction change in body weight across treatment arms at 24 weeks, defined as absolute body weight change.
To assess the impact of pitavastatin vs. rosuvastatin/ezetimibe on low-density lipoproteins (LDL) concentration | 24 weeks
  Mean change in LDL as absolute change from baseline to 24 weeks across treatment arms

SECONDARY OUTCOMES:
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on body mass index (BMI )- weight and height will be combined to report BMI in kg/m^2 | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on waist (cm) to hip (cm) ratio | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on waist (cm) to height (cm) ratio | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on systolic and diastolic blood pressure (mm Hg) | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on Atherosclerotic cardiovascular disease risk score (ASCVD) - calculation of a person's10-year risk (%) of having a cardiovascular problem. | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on fasting lipids including: Total Cholesterol (mmol/L), LDL (mmol/L), High-Density Lipoproteins (HDL) (mmol/L), Triglycerides (mmol/L) | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on fasting glucose (mmol/L) | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on haemoglobin A1C (%) | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on measures of fatty liver disease: Liver Function Tests - Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (U/L), FibroScan (kPa) | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on inflammatory biomarkers (tested centrally on stored research samples) | 48 weeks
To assess the impact of dapagliflozin vs. placebo from baseline to 48 weeks on Serious adverse events. | 48 weeks
To assess the impact of pitavastatin vs. rosuvastatin/ezetimibe from baseline to 48 weeks on fasting lipids including: Total Cholesterol (mmol/L), LDL (mmol/L), High-Density Lipoproteins (HDL) (mmol/L), Triglycerides (mmol/L) | 48 weeks
To assess the impact of pitavastatin vs. rosuvastatin/ezetimibe from baseline to 48 weeks on Atherosclerotic cardiovascular disease risk score (ASCVD) - calculation of a person's10-year risk (%) of having a cardiovascular problem. | 48 weeks
To assess the impact of pitavastatin vs. rosuvastatin/ezetimibe from baseline to 48 weeks on inflammatory biomarkers (tested centrally on stored research samples) | 48 weeks
To assess the impact of pitavastatin vs. rosuvastatin/ezetimibe from baseline to 48 weeks on serious adverse events | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MD, Principal Investigator — Kirby Institute
Locations (10):
- Hospital Ramos Mejía, Buenos Aires, Argentina
- Australia (2):
  - St Vincent's Hospital, Sydney, New South Wales
  - Austin Health, Melbourne, Victoria
- CART-CRS, Chennai, Tamil Nadu, India
- Universiti Malaya Medical Centre, Kuala Lumpur, Malaysia
- Institute of Human Virology, Nigeria, Abuja, Nigeria
- Desmond Tutu Health Foundation, Cape Town, South Africa
- HIV-NAT, Bangkok, Thailand
- Infectious Diseases Institute, Makerere University, Kampala, Uganda
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe